CLINICAL TRIAL: NCT07016399
Title: A Phase II Neoadjuvant Clinical Trial of the Androgen Receptor Inhibitor Darolutamide in Early-Stage Androgen Receptor Positive (AR+) Triple-Negative Breast Cancer
Brief Title: Neoadjuvant Darolutamide Alone or in Combination With Standard Therapy for Stage II-IIIA, AR+, TNBC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vandana Abramson (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Vandana Abramson, Principal Investigator, Vanderbilt-Ingram Cancer Center
Organization: Vanderbilt-Ingram Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICC-VCBRE23490; NCI-2025-03600 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VICC-VCBRE23490 (Other: Vanderbilt University/Ingram Cancer Center); P30CA068485 (NIH)
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Triple-Negative Breast Carcinoma
Keywords: Androgen Receptor-Positive; Luminal Androgen Receptor
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Specimen Handling; Carboplatin; Cyclophosphamide; darolutamide; Doxorubicin; Epirubicin; depelestat; Magnetic Resonance Spectroscopy; Paclitaxel; Taxes; pembrolizumab; Surgical Procedures, Operative; High-Energy Shock Waves

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Standard chemotherapy + immunotherapy) (Active Comparator): Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle, paclitaxel IV on days 1, 8, and 15 of each cycle, and carboplatin IV on days 1, 8, and 15 of each cycle. Cycles repeat every 21 days for up to 4 cycles (cycles 1-4) in the absence of disease progression or unacceptable toxicity. Then, patients receive pembrolizumab IV over 30 minutes, cyclophosphamide IV, and doxorubicin IV or epirubicin IV on day 1 of subsequent cycles. Cycles repeat every 21 days for up to an additional 4 cycles (cycles 5-8) in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo surgery on study, as well as US or MRI, blood sample collection, and breast biopsies throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Breast Biopsy Procedure; Drug: Carboplatin; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Epirubicin; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Biological: Pembrolizumab; Procedure: Surgical Procedure; Procedure: Ultrasound Imaging
- Arm B (Standard chemotherapy + immunotherapy + darolutamide) (Experimental): Patients receive darolutamide PO BID for 14 days in the absence of disease progression or unacceptable toxicity. Patients then receive darolutamide PO BID, pembrolizumab IV over 30 minutes on day 1 of each cycle, and paclitaxel IV on days 1, 8, and 15 of each cycle, and carboplatin IV on days 1, 8, and 15 of each cycle. Cycles repeat every 21 days for up to 4 cycles (cycles 1-4) in the absence of disease progression or unacceptable toxicity. Then, patients receive pembrolizumab IV over 30 minutes, cyclophosphamide IV, and doxorubicin IV or epirubicin IV on day 1 of subsequent cycles. Cycles repeat every 21 days for up to an additional 4 cycles (cycles 5-8) in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo surgery on study, as well as US or MRI, blood sample collection, and breast biopsies throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Breast Biopsy Procedure; Drug: Carboplatin; Drug: Cyclophosphamide; Drug: Darolutamide; Drug: Doxorubicin; Drug: Epirubicin; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Biological: Pembrolizumab; Procedure: Surgical Procedure; Procedure: Ultrasound Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Breast Biopsy Procedure — Undergo breast biopsies
  Other Names: Breast Biopsy
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Darolutamide — Given PO
  Other Names: Antiandrogen ODM-201; BAY 1841788; BAY-1841788; BAY1841788; Nubeqa; ODM 201; ODM-201; ODM201
  Arms: Arm B (Standard chemotherapy + immunotherapy + darolutamide)
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Epirubicin — Given IV
  Other Names: 4'-epi DX; 4'-Epiadriamycin; 4'-Epidoxorubicin; Epi DX; Epidoxorubicin; Pidorubicin
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
Procedure: Surgical Procedure — Undergo breast surgery
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery
Procedure: Ultrasound Imaging — Undergo US
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; Ultrasound; Ultrasound Test; Ultrasound, Medical; US

SUMMARY:
This phase II trial compares the effect of adding darolutamide to standard therapy versus standard therapy alone before surgery for the treatment of patients with stage II-IIIA androgen receptor positive triple-negative breast carcinoma. Standard therapy before surgery for triple-negative breast cancer typically consists of a combination of chemotherapy and immunotherapy drugs. Chemotherapy drugs, such as carboplatin, paclitaxel, doxorubicin and cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Darolutamide is in a class of medications called androgen receptor inhibitors. It works by blocking the effects of androgen (a male reproductive hormone) to stop the growth and spread of tumor cells. Giving darolutamide in combination with standard therapy before surgery may make the tumor smaller and may reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the mean ΔKi-67 level between the darolutamide therapy arm and the control arm.

SECONDARY OBJECTIVES:

I. To determine the pathologic complete response rate (pCR) and overall response rate (ORR) in patients on the darolutamide and control arms.

II. To determine event-free survival (EFS) in patients with androgen receptor positive (AR+) breast cancer in both arms.

III. To correlate the change in Ki-67 at 2 weeks and 6 months with pCR rates and EFS in patients with AR+ breast cancer in both arms.

IV. To monitor circulating tumor deoxyribonucleic acid (ctDNA) throughout treatment and correlate with response in both arms.

V. To correlate percent of nuclear AR positivity with pCR and EFS in both arms.

EXPLORATORY OBJECTIVES:

I. To determine if patients with triple-negative breast cancer (TNBC) experience changes in ctDNA levels while undergoing neoadjuvant therapy.

II. To assess if changes in ctDNA levels correlate with response to neoadjuvant therapy observed in breast cancer tissue biopsies/surgical specimens.

III. To identify AR amplification and ligand binding mutations by whole exome sequencing and evaluate AR transcription targets and AR splice variants by ribonucleic acid sequencing (RNAseq) in baseline, week 2 and residual disease of patients on the darolutamide arm.

IV. To evaluate cell populations and AR transcriptional activity by single-cell RNAseq (scRNAseq) using baseline, week-2 biopsies and residual disease from patients on the darolutamide arm.

V. To assess tumor microenvironment changes in hormone receptors and immune cell populations by multiple immunofluorescences using the CO-Detection by indEXing (CODEX) platform.

VI. To evaluate AR-independent mechanisms of resistance to AR inhibitors using in vitro models for the discovery phase and human tissue for validation studies.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 of each cycle, paclitaxel IV on days 1, 8, and 15 of each cycle, and carboplatin IV on days 1, 8, and 15 of each cycle. Cycles repeat every 21 days for up to 4 cycles (cycles 1-4) in the absence of disease progression or unacceptable toxicity. Then, patients receive pembrolizumab IV over 30 minutes, cyclophosphamide IV, and doxorubicin IV or epirubicin IV on day 1 of subsequent cycles. Cycles repeat every 21 days for up to an additional 4 cycles (cycles 5-8) in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo surgery on study, as well as ultrasound (US) or magnetic resonance imaging (MRI), blood sample collection, and breast biopsies throughout the study.

ARM B: Patients receive darolutamide orally (PO) twice daily (BID) for 14 days in the absence of disease progression or unacceptable toxicity. Patients then receive darolutamide PO BID, pembrolizumab IV over 30 minutes on day 1 of each cycle, and paclitaxel IV on days 1, 8, and 15 of each cycle, and carboplatin IV on days 1, 8, and 15 of each cycle. Cycles repeat every 21 days for up to 4 cycles (cycles 1-4) in the absence of disease progression or unacceptable toxicity. Then, patients receive pembrolizumab IV over 30 minutes, cyclophosphamide IV, and doxorubicin IV or epirubicin IV on day 1 of subsequent cycles. Cycles repeat every 21 days for up to an additional 4 cycles (cycles 5-8) in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo surgery on study, as well as US or MRI, blood sample collection, and breast biopsies throughout the study.

After completion of study treatment, patients are followed up after 30-37 days, at 6 months, 12 months, then yearly for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent as well as the ability to understand and the willingness to sign written consent prior to study registration
* Male or female ≥ 18 years of age on the day of signing informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically confirmed newly diagnosed breast cancer with the following requirements:

  * <10% staining for estrogen receptor (ER) and progesterone receptor (PR) by immunohistochemistry (IHC)
  * HER2 negative by fluorescence in situ hybridization (FISH)
  * AR positive: defined as ≥ 80% staining for AR by IHC
* Primary tumor clinically or radiographically ≥ 1cm in size or stage II-IIIA and eligible for neoadjuvant treatment
* Absolute neutrophil count (ANC) ≥ 1500/µL (≤ 28 days prior to first dose of protocol-indicated treatment)
* Platelets ≥ 100,000/µL (≤ 28 days prior to first dose of protocol-indicated treatment)
* Hemoglobin ≥ 9.0 g/dL or ≥ 5.6 mmol/L (≤ 28 days prior to first dose of protocol-indicated treatment)
* Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min (as calculated by the Cockcroft-Gault Formula or calculated/measured by an alternative established institutional standard consistently applied across participants at the site) (≤ 28 days prior to first dose of protocol-indicated treatment)
* Total bilirubin ≤ 1.5 times institutional upper limit of normal (ULN), or direct bilirubin ≤ ULN for participants with total bilirubin > 1.5 x ULN (≤ 28 days prior to first dose of protocol-indicated treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 times institutional upper limit of normal (ULN) (≤ 28 days prior to first dose of protocol-indicated treatment)
* Calcium ≤ 11.5 mg/dL or ≤ 2.9 mmol/L; in patients with albumin outside the normal range, calcium (corrected for albumin) must be ≤ 11.5 mg/dL or ≤ 2.9 mmol/L (≤ 28 days prior to first dose of protocol-indicated treatment)
* Women must not be breastfeeding and further agree to not breastfeed during study treatment and for at least 120 days after completion of treatment
* A woman of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test during screening within 21 days prior to receiving first dose of protocol-indicated treatment, and must agree to follow instructions for using acceptable contraception from the time of signing consent, and until at least 120 days after completion of treatment
* Men must refrain from donating sperm for at least 120 days after completion of treatment
* A man able to father children who is sexually active with a WOCBP must agree to follow instructions for using acceptable contraception, from the time of signing consent, and until at least 120 days after completion of treatment

Exclusion Criteria:

* Non-resectable breast cancer as assessed by the primary treating surgeon or evidence of metastatic disease
* Malignancies other than TNBC within 5 years prior to randomization, with the exception of those with a negligible risk of metastases or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer)
* Patient is pregnant or breastfeeding
* Patients with moderate hepatic impairment (Child-Pugh Class B cirrhosis or higher)
* Is currently participating in or within four weeks prior to receiving first dose of study treatment in a study of an investigational agent or investigational device

  * Participants who have entered the follow-up phase of an investigational study may participate as long as it has been four weeks after the last dose or last exposure to the previous investigational agent or investigational device
* Recipient of previous allogeneic tissue/solid organ transplant
* Known severe hypersensitivity (≥ Grade 3) to study drug, pembrolizumab, carboplatin, doxorubicin/epirubicin, paclitaxel, or cyclophosphamide and/or any of the excipients of these drugs
* History of myocarditis or pericarditis or other known underlying heart disease that is clinically significant by investigator judgment (for example, cardiomyopathy, congestive heart failure with New York Heart Association [NYHA] functional classification III or IV, symptomatic arrhythmia not controlled by medication, unstable angina, history of acute myocardial infarction). History of cerebrovascular accident (including transient ischemic attack [TIA]) within the past six months (24 weeks) prior to starting study treatment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection/sepsis, or psychiatric illness/social situations that would limit compliance with study requirements
* Known conditions that would preclude the use of checkpoint inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2033-10 (Estimated)

PRIMARY OUTCOMES:
Mean ΔKi-67 level | Baseline up to 5 years
  The two-sample t-test as well as the Wilcoxon Rank-Sum test will be applied to examine the magnitude of ΔKi-67 between the two study arms. The 95% confidence interval (CI) of the mean difference of ΔKi-67 level between two treatment arms will be reported.

SECONDARY OUTCOMES:
Association between ΔKi-67 level and pathologic complete response rate (pCR) status | Baseline up to 5 years
  The exact 95% CIs for pCR will be reported. The generalized linear model will be used to study the correlation between changes of the Ki-67 level and pCR status. In addition, the generalized linear model will be applied to test the correlation between post treatment Ki-67 level and pCR status.
Overall response rate (ORR) | From registration to disease progression or death due to any cause, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method with 95% CIs.
Event-free survival (EFS) | From registration to disease progression or death due to any cause, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method with 95% CIs. The CI based on the Greenwood's variance will be reported. In addition, the two treatment arms as well as the possible risk factors will be compared for survival using the log-rank test. For the multivariable analysis, the proportional hazards Cox model will be applied to investigate potential prognostic factors, such as age of disease onset, on the survival data. The adjusted p-values of the odds ratios and the adjusted 95% CI will be reported.
Correlation of change in Ki-67 with pCR rates and EFS | At 2 weeks and 6 months
  The exact 95% CIs for pCR will be reported. The generalized linear model will be used to study the correlation between changes of the Ki-67 level and pCR status. In addition, the investigators will apply the generalized linear model to test the correlation between post treatment Ki-67 level and pCR status. The study survival will be estimated using the Kaplan-Meier method with 95% CIs. The CI based on the Greenwood's variance will be reported.
Monitor circulating tumor DNA throughout study to correlate with disease response | Baseline up to 5 years
  To assess if changes in ctDNA levels correlate with response to neoadjuvant therapy observed in breast cancer tissue biopsies/surgical specimens
Correlation of percentage of nuclear androgen receptor positivity with pCR and EFS | Baseline up to 5 years
  Will be estimated using the Kaplan-Meier method with 95% CIs.

CONTACTS AND LOCATIONS:
Overall Officials: Vandana G Abramson, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (1):
- Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee, United States